CLINICAL TRIAL: NCT05215041
Title: To Study the Effectiveness and Safety of the Trail of Labor in Full Term Pregnant Women With Cesarean Section After Spontaneous Labor: a Multi-center, Prospective, Observational Study
Brief Title: The Effectiveness and Safety of the Trial of Labor in Full Term Pregnant Women With Cesarean Section After Spontaneous Labor
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: JPPTOLAC-03
Record Dates: First submitted 2021-12-30; First posted 2022-01-31 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Trial of Labor After Cesarean; Vaginal Birth After Cesarean; Spontaneous Labor

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cesarean section group
  Interventions: Other: Non intervention
- Non-cesarean section group
  Interventions: Other: Non intervention

INTERVENTIONS:
Other: Non intervention — If the vaginal delivery is failed after spontaneous labor for up to 24h, they will receive cesarean section

SUMMARY:
This study is a multi-center, prospective, observational clinical trial study. 510 full-term pregnant women will be enrolled as subjects, and the ratio of eligible subjects in the two groups is 1:1. In the cesarean section group, full term pregnant women with one prior cesarean section after spontaneous labor who are willing to try the trial of labor after cesarean (TOLAC) and in accordance with the criteria according to the 2016 China vaginal birth after cesarean (VBAC) clinical management guidelines will be enrolled and recorded by our homemade registration form of TOLAC. In the non-cesarean section group, pregnant women after 37 weeks of gestation after spontaneous labor but without vaginal labor contraindications will be enrolled. After spontaneous labor for 24h, their final delivery mode will be recorded. In the following 42 days postpartum, their complications and the neonatal outcome will be followed up.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers sign the informed consent
2. Age: 20-40 years;
3. Singleton, a cephalic presentation;
4. No contradiction to vaginal delivery; 5.39~42 weeks; 6.Spontaneous labor

Exclusion criteria:

1. Konwn contraindication to vaginal delivery or severe complications;
2. Multiple gestation;
3. Uterine malformation;
4. Severe psychiatric disorder;
5. Without family's support.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: In the cesarean section group, the extra inclusion criteria includes: Only one prior low transverse uterine incision;Extra exclusion criteria:1. With mutiple history of c esction;2. Prior extensive transfundal uterine surgery, such as for fetal surgery, myomectomy, or uterine reconstruction; Prior classical vertical uterine incision, or an inverted "T" or "J" incision;3. Short interpregnancy interval;4.Prior uterine rupture or dehiscence, or cesarean scar pregnancy;4.Evaluated fetal birth weight> 4000 g.
  In the non-cesarean section group, the extra criteria should include: nulliparous
Sampling Method: Probability Sample
Enrollment: 510 (Estimated)
Dates: Start 2022-01-28 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Vignial birth rate | 24 hours
  After spontaneous labor for up tp 24h, the mode of delivery will be konwn and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Jiang Ziyan, Ph.D, Principal Investigator — Department of Obstetrics and Gynecology, First Affiliated Hospital of Nanjing Medical University
Locations (1):
- First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lassey SC, Robinson JN, Kaimal AJ, Little SE. Outcomes of Spontaneous Labor in Women Undergoing Trial of Labor after Cesarean as Compared with Nulliparous Women: A Retrospective Cohort Study. Am J Perinatol. 2018 Jul;35(9):852-857. doi: 10.1055/s-0037-1619448. Epub 2018 Jan 24. PMID 29365328
- [Background] Al-Shaikh G, Al-Mandeel H. The outcomes of trial of labour after cesarean section following induction of labour compared to spontaneous labour. Arch Gynecol Obstet. 2013 Jun;287(6):1099-103. doi: 10.1007/s00404-013-2709-z. Epub 2013 Jan 11. PMID 23307166